CLINICAL TRIAL: NCT04870528
Title: Adjunctive Effect of Pulsed Electromagnetic Field on Quadriceps Muscle Strength After Burn Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walaa Abd Elaziem Abd Elaziz (Other)
Responsible Party: Sponsor-Investigator, Walaa Abd Elaziem Abd Elaziz, Assistant lecturer of physical therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/002906
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Lower Limb Burn

STUDY DESIGN:
Intervention Model Description: In this study, the patients will be assigned into two equal groups :
  study group which will receive (Pulsed Electromagnetic Field therapy and quadriceps strengthening exercises), control group which will receive (Quadriceps strengthening exercises).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants are suffering from lower limb burn with second-degree burn ( Partial thickness of thermal injury) and total body surface area (TBSA) from 20% to 35%.The care provider are burn center stuff. The investigator is a physical therapist(myself).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): - This group will be composed of 30 patients with lower limb burn of second-degree. Subjects will receive pulsed magnetic field over thigh areas for 24 sessions over a period of 8 weeks (3sessions/week) with receiving strengthening exercises for quadriceps muscle and traditional physical therapy program in the form of range of motion exercise, stretching, splinting, massage, functional training for ambulation and activities of daily living.
  Interventions: Device: pulsed electromagnetic field device; Other: Free weights for Strengthening Exercise
- control group (Active Comparator): Subjects will receive strengthening exercises for quadriceps muscle and traditional physical therapy program in the form of range of motion exercise, stretching, splinting, massage, functional training for ambulation and activities of daily living for 24 sessions over a period of 8 weeks (3sessions/week)
  Interventions: Other: Free weights for Strengthening Exercise

INTERVENTIONS:
Device: pulsed electromagnetic field device — the pulsed electromagnetic field device treatment parameters will be set as 15 Hz frequency, 20 gauss amplitude, and 20 minutes as total treatment duration.
  Arms: Experimental group
Other: Free weights for Strengthening Exercise — • Parameters of the exercise program: Intensity : The weight or load the patients lifted is set at 50-60% of their individual 1RM , 3 sets of 10 repetitions during the first week. During the second week, the lifting load is increased to 70-75% (3 sets of 10 repetitions) of their individual 1RM and continued for weeks 2-6. After this, training intensity is increased to 80-85% of the 1 RM and implemented from weeks 7-8.
  Frequency: 3 sessions per week for 8 weeks. Number of repetitions: 3 sets,10 repetitions in each set. Total treatment duration: 8 weeks

SUMMARY:
The aim of this study is to examine whether Pulsed Electromagnetic Field therapy combined with strengthening exercises will have a positive effect on quadriceps muscle strength in lower limb burn .

DETAILED DESCRIPTION:
• Subjects: Sixty patients with lower limb burn, subdivided into two groups each one has 30 patients.

* Group (A) = Pulsed Electromagnetic Field therapy and quadriceps strengthening exercises group.
* Group (B) = quadriceps strengthening exercises group. • Equipment and tools:

  1. Measurements tools:

     Isokinetic dynamometer : to measure the quadriceps muscle peak torque before the treatment and after 8 weeks of treatment for both groups.
  2. Therapeutic tools:

Pulsed Electromagnetic Field therapy device and free weights for strengthening of quadriceps muscle.

ELIGIBILITY:
Inclusion Criteria:

* - Patients are males.
* Their age will range from (25-40) years.
* Patients will suffer from second-degree burn ( Partial thickness of thermal injury).
* Total body surface area (TBSA) for the burns will be ranged from 20% to 35% .
* They will be selected from Outpatient Clinic of Faculty of Physical Therapy and Burn Unit at Om El-Obour Hospital.
* Patients will begin the training program after complete wound healing.
* All patients will receive traditional physical therapy program in the form of range of motion exercise, stretching, splinting, massage, functional training for ambulation and activities of daily living.
* Patients will be given their informed consent.

Exclusion Criteria:

* - Patients who participate in any rehabilitation program to improve muscle strength prior to the study.
* Musculoskeletal disorders that will impair performance during training and tests.
* Equilibrium disorders.
* Uncontrolled cardiovascular or pulmonary diseases .
* Neurological and renal disorders.
* metabolic or vascular disease with a neurological component such as diabetes,
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders.
* Subjects with burn to the posterior thigh with knee flexion contracture, which affected the function of the quadriceps muscle.
* Lower limb lymphedema or lipoedema.
* Athletic subjects.
* Subjects with morbid obesity.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Isokinetic dynamometer for measuring The peak torque of the quadriceps muscle | 8 weeks
  * Patients will warm up for 5 min on a cycle ergometer then quadriceps, hamstrings and calf muscles will be stretched 3 times with a 30 seconds stretch and a 30 seconds rest.
  * Patients will be positioned in an isokinetic dynamometer. The measurements are carried out with the backrest reclined 5° from vertical and knees flexed 90 degrees and straps fixing the trunk, waist and distal thigh. The rotation axis of the dynamometer is aligned with the axis of the knee joint at the level of the lateral epicondyle of the femur while it is attached to the distal part of the leg about 5cm above the medial malleolus and isokinetic test is performed at angular velocity of 150 degree per second.
  * For familiarization, Patients will perform a series of three submaximal contractions. After warming up, subjects are requested to perform ten maximal voluntary contractions consecutively without rest in between.
  * There will be three minutes of resting before repeating the test

CONTACTS AND LOCATIONS:
Overall Officials: Walaa A Elaziz, master, Principal Investigator — lecturer assistant at faculty of physical therapy, Cairo University
Locations (1):
- Cairo University, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No